CLINICAL TRIAL: NCT05798286
Title: Does Bedside Ultrasound Clot Elasticity Measurement Reduce Intraoperative Transfusion During Double-lung Transplantation?
Brief Title: Quantra® System With the QPlus® Cartridge in Double-lung Transplantation
Acronym: QUANTRANS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2020_0084
Record Dates: First submitted 2023-03-16; First posted 2023-04-04 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Lung Diseases; Transplant-Related Disorder
Keywords: Resonance sonorheometry; Viscoelastic testing; Quantra system; Lung transplantation
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QUANTRA group (Experimental): Adult subjects (18 years-old or older) undergoing double-lung transplantation: transfusion algorithm based on whole blood viscoelastic test with Quantra® + standard coagulation test. These samples are collected at five standard surgical time points:
  * on arrival at the hospital on the day of surgery,
  * after first pulmonary artery clamping,
  * after first graft implantation,
  * after second graft implantation,
  * at end-surgery status.
  Interventions: Other: Quantra
- Control group (Active Comparator): Adult subjects (18 years-old or older) undergoing double-lung transplantation: standard transfusion algorithm based on standard practice and coagulation test. These samples are collected at five standard surgical time points:
  * on arrival at the hospital on the day of surgery,
  * after first pulmonary artery clamping,
  * after first graft implantation,
  * after second graft implantation,
  * at end-surgery status.
  Interventions: Other: Control

INTERVENTIONS:
Other: Quantra — The study plans to collect 2 additional 3 mL citrate tubes of venous blood in addition to the platelet and blood counts.
  Arms: QUANTRA group
Other: Control — The study plans to collect 1 additional 3 mL citrate tubes of venous blood in addition to the platelet and blood counts at each time.
  Arms: Control group

SUMMARY:
Transfusion in lung transplantation is common, and despite improved techniques and limitations in the use of mechanical circulatory support (MCS), the incidence of massive transfusion has remained stable over the years. The consequences of blood transfusion (blood cells, plasma, platelet concentrates) are deleterious for patients and increase primary graft dysfunction and mortality risk.

Whole blood viscoelastic testing devices have shown its effectiveness in monitoring coagulation and fibrinolytic function during cardiac surgery, liver transplantation or trauma. So far, few delocalized biology tools have been evaluated in lung transplantation.

The main objective of this study is to determine if the use of a transfusion algorithm based on whole blood viscoelastic test with Quantra® test reduce transfusion during lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing double-lung transplantation
* Patient is ≥ 18 years-old
* Patient is willing to participate, and is willing to consent
* Patient affiliated to a national health insurance

Exclusion Criteria:

* Patient is younger than 18 years-old
* Patient with an indication for non double-lung transplantation
* Patient under extracorporeal membrane oxygenation in bridge to transplantation
* Patient with surgery under cardiopulmonary bypass
* Patient benefiting from a multi-organ transplantation
* Patient being deprived of liberty or under guardianship
* Patient refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2025-10-03 (Estimated)

PRIMARY OUTCOMES:
Labile blood products measure | 24 hours
  Number of labile blood products (red blood cells pack + fresh frozen plasma) transfused in the operating room.

SECONDARY OUTCOMES:
The impact of Quantra® on the administration of each type of transfusion during surgery and within 24 hours after transplantation | 24 hours
  Number of patients receiving each type of labile blood product and the number of red blood cell pack, platelet concentrates, fresh frozen plasma, and fibrinogen administered during surgery and within 24 hours following surgery
blood loss during surgery | 24 hours
  volume of blood lost during surgery.
The occurrence of acute primary graft dysfunction at day 3. | 3 days
  Grade 3 primary graft dysfunction measured on the 3rd postoperative day
Quality of life six months after surgery using EQ-5D-5L questionnaire including five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression | 6 months
  Quality of life questionnaire assement using the EuroQol Group's five-level EuroQol five-dimensional questionnaire (EQ-5D-5L) including five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Hospital mortality, at 30 days, 90 days, and 12 months | 12 months
  Hospital mortality rate, at 30 days, 90 days, and at 12 months.
Number of transfused labile blood products during the length of an individual's stay in hospital | up to 12 months
  The number of transfused labile blood products will evaluated during the length of an individual's stay in hospital
Duration of stay in intensive care | up to 12 months
  The duration of stay in intensive care will evaluated during the length of an individual's stay in hospital
The median cost of transfused labile blood products | up to 12 months
  The median cost of transfused labile blood products will evaluated during the length of an individual's stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Julien Fessler, MD, Study Director — Foch Hospital; Tiffany Pascreau, MD, Principal Investigator — Foch Hospital
Locations (1):
- Foch Hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Triulzi DJ, Griffith BP. Blood usage in lung transplantation. Transfusion. 1998 Jan;38(1):12-5. doi: 10.1046/j.1537-2995.1998.38198141492.x. PMID 9482388
- [Background] Cernak V, Oude Lansink-Hartgring A, van den Heuvel ER, Verschuuren EAM, van der Bij W, Scheeren TWL, Engels GE, de Geus AF, Erasmus ME, de Vries AJ. Incidence of Massive Transfusion and Overall Transfusion Requirements During Lung Transplantation Over a 25-Year Period. J Cardiothorac Vasc Anesth. 2019 Sep;33(9):2478-2486. doi: 10.1053/j.jvca.2019.03.060. Epub 2019 Mar 30. PMID 31147209
- [Background] Huddleston SJ, Jackson S, Kane K, Lemke N, Shaffer AW, Soule M, Hertz M, Shumway S, Qi S, Perry T, Kelly R. Separate Effect of Perioperative Recombinant Human Factor VIIa Administration and Packed Red Blood Cell Transfusions on Midterm Survival in Lung Transplantation Recipients. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):3013-3020. doi: 10.1053/j.jvca.2020.05.038. Epub 2020 Jun 3. PMID 32718888
- [Background] Seay T, Guinn N, Maisonave Y, Fuller M, Poisson J, Pollak A, Bryner B, Haney J, Klapper J, Hartwig M, Bottiger B. The Association of Increased FFP:RBC Transfusion Ratio to Primary Graft Dysfunction in Bleeding Lung Transplantation Patients. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):3024-3032. doi: 10.1053/j.jvca.2020.05.043. Epub 2020 Jun 7. PMID 32622711
- [Background] Cimic N, Tulleken JE, Zijlstra JG, van der Bij W, Boonstra PW. Recombinant factor VIIa for refractory hemorrhage after lung transplantation. Transplantation. 2005 Mar 27;79(6):741-2. doi: 10.1097/01.tp.0000147319.66838.71. No abstract available. PMID 15785389
- [Background] Felten ML, Fischler M. Intraoperative use of activated recombinant factor VII for refractory bleeding in complicated lung transplantations. J Cardiothorac Vasc Anesth. 2010 Apr;24(2):382-3. doi: 10.1053/j.jvca.2009.06.006. Epub 2009 Aug 19. No abstract available. PMID 19695905
- [Background] Detterbeck FC, Egan TM, Mill MR. Lung transplantation after previous thoracic surgical procedures. Ann Thorac Surg. 1995 Jul;60(1):139-43. PMID 7598576
- [Background] Ius F, Kuehn C, Tudorache I, Sommer W, Avsar M, Boethig D, Fuehner T, Gottlieb J, Hoeper M, Haverich A, Warnecke G. Lung transplantation on cardiopulmonary support: venoarterial extracorporeal membrane oxygenation outperformed cardiopulmonary bypass. J Thorac Cardiovasc Surg. 2012 Dec;144(6):1510-6. doi: 10.1016/j.jtcvs.2012.07.095. Epub 2012 Aug 31. PMID 22944092
- [Background] Hoechter DJ, Shen YM, Kammerer T, Gunther S, Weig T, Schramm R, Hagl C, Born F, Meiser B, Preissler G, Winter H, Czerner S, Zwissler B, Mansmann UU, von Dossow V. Extracorporeal Circulation During Lung Transplantation Procedures: A Meta-Analysis. ASAIO J. 2017 Sep/Oct;63(5):551-561. doi: 10.1097/MAT.0000000000000549. PMID 28257296
- [Background] Adelmann D, Koch S, Menger J, Opfermann P, Jaksch P, Hoetzenecker K, Kurz M, Mouhieddine M, Steinlechner B. Risk factors for early bleeding complications after lung transplantation - a retrospective cohort study. Transpl Int. 2019 Dec;32(12):1313-1321. doi: 10.1111/tri.13491. Epub 2019 Aug 30. PMID 31402529
- [Background] Kesten S, de Hoyas A, Chaparro C, Westney G, Winton T, Maurer JR. Aprotinin reduces blood loss in lung transplant recipients. Ann Thorac Surg. 1995 Apr;59(4):877-9. doi: 10.1016/0003-4975(95)00051-l. PMID 7535041
- [Background] Balsara KR, Morozowich ST, Lin SS, Davis RD, Phillips-Bute BG, Hartwig M, Appel JZ, Welsby IJ. Aprotinin's effect on blood product transfusion in off-pump bilateral lung transplantation. Interact Cardiovasc Thorac Surg. 2009 Jan;8(1):45-8. doi: 10.1510/icvts.2008.178749. Epub 2008 Jul 31. PMID 18669527
- [Background] Bittner HB, Richter M, Kuntze T, Rahmel A, Dahlberg P, Hertz M, Mohr FW. Aprotinin decreases reperfusion injury and allograft dysfunction in clinical lung transplantation. Eur J Cardiothorac Surg. 2006 Feb;29(2):210-5. doi: 10.1016/j.ejcts.2005.12.001. PMID 16386921
- [Background] Bittner HB, Binner C, Dahlberg P, Mohr FW. Reducing ischemia-reperfusion injury in clinical lung transplantation. Transplant Proc. 2007 Mar;39(2):489-92. doi: 10.1016/j.transproceed.2006.12.005. PMID 17362765
- [Background] Marasco SF, Pilcher D, Oto T, Chang W, Griffiths A, Pellegrino V, Chan J, Bailey M. Aprotinin in lung transplantation is associated with an increased incidence of primary graft dysfunction. Eur J Cardiothorac Surg. 2010 Feb;37(2):420-5. doi: 10.1016/j.ejcts.2009.08.007. Epub 2009 Sep 19. PMID 19767212
- [Background] Herrington CS, Prekker ME, Arrington AK, Susanto D, Baltzell JW, Studenski LL, Radosevich DM, Kelly RF, Shumway SJ, Hertz MI, Bittner HB, Dahlberg PS. A randomized, placebo-controlled trial of aprotinin to reduce primary graft dysfunction following lung transplantation. Clin Transplant. 2011 Jan-Feb;25(1):90-6. doi: 10.1111/j.1399-0012.2010.01319.x. Epub 2010 Aug 19. PMID 20731686